CLINICAL TRIAL: NCT01722188
Title: Optim Lead Insulation Material Registry
Brief Title: Lead Registry for Optim Leads
Acronym: OPTIMUM
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: CD0196
Record Dates: First submitted 2012-11-02; First posted 2012-11-06 (Estimated); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Optim Lead Insulation Related Adverse Events
Keywords: Optim; Insulation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Optim Leads

SUMMARY:
This is a prospective, multi-center, actively monitored, long term data collection registry. Any Patient that receives a market released St. Jude Medical (SJM) Optim lead and a compatible market released cardia rhythm management (CRM) implantable pulse generator is eligible for enrollment into the registry.

DETAILED DESCRIPTION:
Patients are enrolled in the registry up to 180 days post implantation of an Optim lead. Patients with Optim™ ICD leads and Quicksite®/Quickflex®/Quickflex® µ/Quartet® LV leads are followed indefinitely following enrollment. Patients with other Optim leads are followed for a period of 60 months after Optim™ lead implantation. The follow-up plan for this registry is based on the established follow-up practices currently used by each of the respective registry centers. Patients are followed according to the center's standard follow-up schedule.

At each office/clinic follow-up visit standard electrical measurements are collected. During system revision in a patient with either Optim™ ICD leads, Quicksite®, Quickflex®, Quickflex® µ or Quartet® LV lead, cinefluoroscopy (AP, LAO 45° or the best possible LAO view, RAO 45° or the best possible RAO view) should be performed at specific study sites. If cinefluoroscopy or chest X-ray is performed according to the site's standard of care then copies of those should be submitted.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a standard indication for a CRM implantable pulse generator.
* Patient receives a market released SJM Optim lead at implant.
* Patient receives a market released CRM implantable pulse generator at implant.
* Patient is willing to provide authorization for registry participation.
* Complete device implant information, including any Optim lead related adverse event is available

Exclusion Criteria:

* Patient has medical conditions or related factors that would prevent or limit participation (including mechanical tricuspid valves, tricuspid valvular disease, and candidacy for heart transplants within 6 months).
* Patient is < 18 years of age.
* Patient has a life expectancy of < 2 years (malignancies)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients implanted with market released SJM Optim lead and a compatible market released CRM implantable pulse generator (pacemaker, implantable cardioverter defibrillator (ICD), or cardiac resynchronization therapy device (CRT)) is eligible for enrollment into the registry.
Sampling Method: Probability Sample
Enrollment: 14124 (Actual)
Dates: Start 2006-08 (Actual); Primary Completion 2020-07 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Survival from insulation related adverse events | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Grant Kim, Study Director — Abbott Medical Devices
Locations (261):
- United States (245):
  - Heart South Cardiovascular Group PC, Alabaster, Alabama
  - Appalachian Cardiovascular Associates, Fort Payne, Alabama
  - North Alabama Cardiology Center, Gadsden, Alabama
  - Cardiology Associates of Mobile, Inc., Mobile, Alabama
  - Alaska Heart Institute, Anchorage, Alaska
  - Pima Heart Physicians, PC, Tucson, Arizona
  - Southern Arizona VA Health Care System, Tucson, Arizona
  - Arkansas Cardiology, Little Rock, Arkansas
  - *Little Rock Cardiology Clinic, Little Rock, Arkansas
  - Northwest Cardiology, Springdale, Arkansas
  - Westside Cardiovascular Associates, Beverly Hills, California
  - Raymond Schaerf, MD, Burbank, California
  - Mills-Peninsula Cardiovascular Specialists, Burlingame, California
  - Center for Interventional Cardiology and Nephrology, Encino, California
  - Cardiac Institute, Fresno, California
  - Mid Valley Cardiology, Fresno, California
  - Cardiac Care Specialists, Glendale, California
  - Glendale Memorial Hospital and Medical Center, Glendale, California
  - Apex Cardiology, Inglewood, California
  - Kartik Thaker, MD Inc., Lakewood, California
  - Omid Vahdat M.D., Los Alamitos, California
  - Donna Gallik MD, Los Angeles, California
  - Jeffrey Goodman MD, Los Angeles, California
  - Payam Yashar M.D., Los Angeles, California
  - Stephen S. Ehrlich, MD, Mission Viejo, California
  - Inland Valley Cardiovascular Center, Murrieta, California
  - Mehrdad Ariani MD, Northridge, California
  - Soltera Yasuda & Associates, Northridge, California
  - Cabrillo Cardiology Medical Group, Oxnard, California
  - Alejandro Garcia MD, Oxnard, California
  - Desert Heart Physicians, Palm Springs, California
  - Southern California Heart Specialists, Pasadena, California
  - William A Stellar, MD, Rancho Mirage, California
  - Cardiac Rhythm Specialists, Inc., Reseda, California
  - Heart Center of Riverside, Riverside, California
  - Mercy Medical Group Cardiology, Sacramento, California
  - Salinas Valley Memorial Hospital, Salinas, California
  - Bruce A. Ourieff MD, Santa Maria, California
  - Sun City Cardiology Medical Center, Incorporated, Sun City, California
  - Sun City Cardiology Medical Center, Inc, Sun City, California
  - Michael Burnam, MD, Tarzana, California
  - Richard P. Cain, MD, Tarzana, California
  - COR Healthcare Medical Associates, Torrance, California
  - Cardiovascular Consultants, Van Nuys, California
  - Arash Vahdat, MD, Van Nuys, California
  - Shiva Heart Center Medical Group, Wildomar, California
  - Feather River Cardiovascular Institute, Yuba City, California
  - Yuba Sutter Medical Clinic, Yuba City, California
  - Penrose St. Francis Cardiology Associates PC, Colorado Springs, Colorado
  - Pikes Peak Cardiology, Colorado Springs, Colorado
  - Harvard Park Medical, Denver, Colorado
  - South Denver Cardiology Associates PC, Littleton, Colorado
  - Grove Hill Medical Center, New Britain, Connecticut
  - Cardiology Associates of Fairfield County, PC, Norwalk, Connecticut
  - Cardiac Arrhythmia Services, Boca Raton, Florida
  - Bradenton Heart Center, Bradenton, Florida
  - Bay Area Cardiology Associates PA, Brandon, Florida
  - Florida Cardiology Group, Brooksville, Florida
  - Pinellas Arrhythmia Associates, Clearwater, Florida
  - Okaloosa Heart and Vascular, Crestview, Florida
  - Cardiology Consultants PA, Daytona Beach, Florida
  - The Cardiology Center, Incorporated, Delray Beach, Florida
  - White-Wilson Medical Center - Fort Walton Beach, Fort Walton Beach, Florida
  - The Cardiac & Vascular Institute Research Foundation, LLC, Gainesville, Florida
  - Shands at the University of Florida, Gainesville, Florida
  - Florida Institute For Cardiovascular Care, Hollywood, Florida
  - Jorge Diaz, M.D., P.A., Lake Mary, Florida
  - Clark & Daughtrey Medical Group, PA, Lakeland, Florida
  - Diagnostic and Interventional Cardiology, Melbourne, Florida
  - Melbourne Internal Medicine Associates, Melbourne, Florida
  - Miami International Cardiology Consultants Inc, Miami Beach, Florida
  - Institute of Cardiovascular Research LLC, Ocala, Florida
  - Ram Vasudevan, MD, FACC, Ocala, Florida
  - Central Florida Heart Center, Ocala, Florida
  - Cardiovascular Interventions, P.A., Orlando, Florida
  - Mid-Florida Cardiology Specialist, Orlando, Florida
  - Cardiology Research Associates, Ormond Beach, Florida
  - Cardio Care Center, Palatka, Florida
  - St. Augustine Cardiology Associates, Saint Augustine, Florida
  - Heart Care Research, Sarasota, Florida
  - Sarasota Heart Center, Sarasota, Florida
  - Sarasota Arrhythmia Institute, Sarasota, Florida
  - Dr. Kalpesh Solanki, Summerfield, Florida
  - Tallahassee Research Institute, Tallahassee, Florida
  - Mazhar Majid, M.D., Tamarac, Florida
  - Heart & Vascular Center of Venice, Venice, Florida
  - Athens Heart Center, Athens, Georgia
  - Piedmont Athens Regional Medical Center, Athens, Georgia
  - St. Mary's, Athens, Georgia
  - Piedmont Heart Institute - Buckhead Location, Atlanta, Georgia
  - Northeast Georgia Heart Foundation, Gainesville, Georgia
  - Gwinnet Consultants in Cardiology, Lawrenceville, Georgia
  - Kennestone Heart Physicians, Marietta, Georgia
  - Harbin Clinic Southeastern Cardiovascular Institute, Rome, Georgia
  - South Georgia Cardiology PC, Valdosta, Georgia
  - Fox Valley Cardiovascular Consultants, Aurora, Illinois
  - Provena Saint Joseph Hospital, Elgin, Illinois
  - MidAmerica Cardiovascular Consultants, Oak Lawn, Illinois
  - Rockford Cardiology Associates, Rockford, Illinois
  - Ohio Valley Heart Care, Evansville, Indiana
  - Saint Margaret Mercy Healthcare Centers, Hammond, Indiana
  - River Cities Cardiology, Jeffersonville, Indiana
  - Medical Consultants, Muncie, Indiana
  - Cardiology Associates of NW Indiana, Munster, Indiana
  - Unitypoint, Des Moines, Iowa
  - Cumberland Cardiology, Ashland, Kentucky
  - Cardiology Associates of Kentucky, Lexington, Kentucky
  - Bluegrass Cardiology, Louisville, Kentucky
  - Baptist Health Medical Group, Inc., Madisonville, Kentucky
  - Alexandria Cardiology Clinic, Alexandria, Louisiana
  - Freedman Memorial Cardiology, Alexandria, Louisiana
  - Our Lady of the Lake Hospital, Baton Rouge, Louisiana
  - Cardiovascular Associates, Covington, Louisiana
  - Covington Cardiovascular Care, Covington, Louisiana
  - St. Tammany Heart and Vascular, Covington, Louisiana
  - Heart and Vascular Institute of LA LLC, Lacombe, Louisiana
  - Mike Mounir MD, Lafayette, Louisiana
  - Cardiovascular Specialists of SWLA, Lake Charles, Louisiana
  - Imperial Health, LLP, Lake Charles, Louisiana
  - Cardiology Center, Marrero, Louisiana
  - Gregory C. Sampognaro Interventional Cardiology, Monroe, Louisiana
  - Cardiology Associates Incorporated, Shreveport, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - National Naval Medical Center, Bethesda, Maryland
  - Cardiac Associates PC, Rockville, Maryland
  - Delmarva Heart, Salisbury, Maryland
  - Peninsula Cardiology Associates, P.A., Salisbury, Maryland
  - Alan Schneider, Silver Spring, Maryland
  - Baystate Medical Practice, Florence, Massachusetts
  - The Cardiovascular Specialists, Hyannis, Massachusetts
  - Fallon Clinic, Worcester, Massachusetts
  - Heart Rhythm Specialists of Central Massachusetts, PC, Worcester, Massachusetts
  - University of Massachusetts Medical Center, Worcester, Massachusetts
  - Cardiology and Arrhythmia Consultants P.C., Birmingham, Michigan
  - Regional Cardiology Associates, PLC, Grand Blanc, Michigan
  - Academic Cardiology Associates, Rochester Hills, Michigan
  - Heart Cardiology Consultants, Southfield, Michigan
  - Grand Traverse Heart Associates, Traverse City, Michigan
  - Lingareddy Devireddy, PC, Warren, Michigan
  - St. Luke's Cardiology Associates, Duluth, Minnesota
  - VA Medical Center Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Medical Center Fairview, Minneapolis, Minnesota
  - Coast Cardiovascular Consultants, Biloxi, Mississippi
  - Coast Cardiology Center, Gulfport, Mississippi
  - Hattiesburg Clinic, Hattiesburg, Mississippi
  - Cardiovascular Consultants of Cape Girardeau Inc, Cape Girardeau, Missouri
  - The Heart Care Group, Florissant, Missouri
  - Cardiovascular Consultants (now St. Luke's), Kansas City, Missouri
  - St. Louis University Hospital, St Louis, Missouri
  - County Cardiology, Inc., St Louis, Missouri
  - The Heart Health Center, St Louis, Missouri
  - St. Louis Cardiology Consultants, St Louis, Missouri
  - Methodist Physicians Clinic-Heart Consultants, Omaha, Nebraska
  - Alegent Creighton Health, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Nevada Cardiology Associates, Las Vegas, Nevada
  - Cooper University Hospital, Camden, New Jersey
  - South Jersey Heart Group, Cherry Hill, New Jersey
  - Hunterdon Cardiovascular Associates, Flemington, New Jersey
  - Hamilton Cardiology Associates, Hamilton, New Jersey
  - Atlantic Health System - Morristown Memorial Hospital, Morristown, New Jersey
  - Monmouth Cardiology Associates, LLC, Ocean City, New Jersey
  - Cardiology Consultants of North Jersey, Wayne, New Jersey
  - New Jersey Cardiology Associates, West Orange, New Jersey
  - New Mexico Heart Institute, Albuquerque, New Mexico
  - Adirondack Cardiology Associates, Glens Falls, New York
  - Long Island Heart Associates, Mineola, New York
  - Cardiac Arrhythmia and Pacemaker Center, Roslyn, New York
  - Wayne Heart Internal Medicine, Goldsboro, North Carolina
  - Piedmont Cardiology Associates, Hickory, North Carolina
  - Wake Heart Associates, Raleigh, North Carolina
  - Sanford Research, Fargo, North Dakota
  - Altru Clinic - Main, Grand Forks, North Dakota
  - City Cardiology Associates, Barberton, Ohio
  - Electrophysiology & Pacing Interventionalists, Columbus, Ohio
  - Electrophysiology and Pacing Interventionalists, Columbus, Ohio
  - University Hospitals Elyria Medical Center, Elyria, Ohio
  - Mercy Hospital Fairfield, Fairfield, Ohio
  - Ohio Institute Of Cardiac Care, Springfield, Ohio
  - Heart Care Cardiology Consultants, Inc., Steubenville, Ohio
  - Riverside Medical of Ohio, Steubenville, Ohio
  - Northwest Ohio Cardiology Consultants, Toledo, Ohio
  - Toledo Clinic, Toledo, Ohio
  - Ohio Heart Institute, Youngstown, Ohio
  - Cardiac Arrhythmia Associates, Youngstown, Ohio
  - Khastgir, Terrance M.D., Oklahoma City, Oklahoma
  - Cardiovascular Consultants, Inc., Tulsa, Oklahoma
  - Abington Medical Specialists, Abington, Pennsylvania
  - SouthWestern Pennsylvania Cardiovascular Associates, Butler, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Dubois Regional Cardiology Associates, Sandy, Pennsylvania
  - Donald Guthrie Foundation for Education and Research, Sayre, Pennsylvania
  - Charleston Cardiology, Charleston, South Carolina
  - Coastal Cardiology, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - South Carolina Heart Center, Columbia, South Carolina
  - Pee Dee Cardiology Associates, PA, Florence, South Carolina
  - Piedmont Cardiology, Greenwood, South Carolina
  - The Chattanooga Heart Institute, Chattanooga, Tennessee
  - Mountain States Medical Group Cardiology, Johnson City, Tennessee
  - East Tennessee Heart Consultants - Knoxville, Knoxville, Tennessee
  - Knoxville Cardiovascular Research Group, LLC, Knoxville, Tennessee
  - Arrhythmia Consultants, P.C., Memphis, Tennessee
  - Heart Rhythm Consultants, Austin, Texas
  - Bay City Cardiology Clinic at Matagorda General Hospital, Bay City, Texas
  - Southeast Texas Cardiology, Beaumont, Texas
  - BCS Heart, LLP, College Station, Texas
  - Dallas Heart Group, Dallas, Texas
  - North Texas Heart Center, Dallas, Texas
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - Cardiology Care Consultants, El Paso, Texas
  - Texas Heart Clinic, PA, Fort Worth, Texas
  - Center for Cardiac Arrhythmias, Houston, Texas
  - EP/Cardiology PA, Houston, Texas
  - Willowbrook Cardiovascular Associates, Houston, Texas
  - Cardiovascular Association, P.L.L.C., Humble, Texas
  - Texas Cardiac Center, Lubbock, Texas
  - Permian Cardiology Associates, Midland, Texas
  - Odessa Heart Institute, P. A., Odessa, Texas
  - Miguel E. Castellanos, MD, Orange, Texas
  - South Texas Cardiovascular Consultants, San Antonio, Texas
  - Cardiology Clinic Of San Antonio Pa, San Antonio, Texas
  - Brooke Army Medical Center, Division of Cardiology, San Antonio, Texas
  - Scott & White Memorial Hospital, Temple, Texas
  - Cardiovascular Associates of East Texas, Tyler, Texas
  - Victoria Heart and Vascular, Victoria, Texas
  - Cardiovascular Associates Ltd, Chesapeake, Virginia
  - The Cardiovascular Group, Fairfax, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Riverside Heart Specialists, Hampton, Virginia
  - Harrisonburg Medical Associations, Inc., Harrisonburg, Virginia
  - Virginia Cardiovascular Specialists, Richmond, Virginia
  - Hunter Holmes McGuire VAMC, Richmond, Virginia
  - Bellevue Cardiology, Bellevue, Washington
  - Overlake Internal Medicine Associates, Bellevue, Washington
  - Kitsap Cardiology Consultants, Bremerton, Washington
  - Skagit Valley Medical Center, Mount Vernon, Washington
  - The Heart Institute at Virginia Mason, Seattle, Washington
  - Sacred Heart Medical Center, Spokane, Washington
  - Kootenai Heart Clinics, Spokane, Washington
  - Franciscan Cardiology Associates, Tacoma, Washington
  - Franciscan Heart & Vascular Associates, Tacoma, Washington
  - Cardiology Associates of Green Bay, Ltd., Green Bay, Wisconsin
  - Dean Foundation, Madison, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
- CHR Citadelle, Liège, Belgium
- Germany (15):
  - Praxis Dr. med. Irtel von Brenndorff, Baden-Baden, Bad-wur
  - Praxis Dr. med. Markert, Gaggenau, Bad-wur
  - Praxis Dr. med. Behroz, Heidelberg, Bad-wur
  - Praxis Dr. med. Thomas Fadgyas, Dortmund, N. RHIN
  - Praxis Dr. med. Bernhardt, Annaberg-Buchholz, Saxony
  - Praxis Dr. Med. Stellmach, Chemnitz, Saxony
  - Praxis Frau Dr. med. Strucks, Nossen, Saxony
  - Klinikum Pirna GmbH Klinik für Innere Medizin II, Pirna, Saxony
  - Kreiskrankenhaus des Bördekreises Krankenhaus 4, Oschersleben, Sxnyanh
  - Kardiologische Gem.-Praxis Dres. med. Bischoff / Lang, Erfurt, Thurgia
  - Helios-Klinikum Erfurt GmbH, Erfurt, Thurgia
  - Asklepios Klinik St. Georg, Hamberg
  - Asklepios Klinik Nord Heidberg-Ochsenzoll, Hamberg
  - Asklepios Klinik Altona, Hamberg
  - Praxis Dr. med. Subin, Hamburg